CLINICAL TRIAL: NCT00186303
Title: Autologous and Allogeneic Peripheral Blood Progenitor (PBPC) Transplantation for Patients With Chronic Lymphocytic Leukemia
Brief Title: Transplantation for Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert Negrin, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMT88; 77066; BMT88; NCT00186303
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Leukemia, Lymphocytic, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Procedure: high dose chemotherapy then autologous hematopoietic cell transplant
Procedure: ablative allogeneic hematopoietic cell transplant

SUMMARY:
To evaluate the role of high dose therapy and autologous or allogeneic hematopoietic cell transplantation for the treatment of chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
To determine effectiveness of allogeneic transplantation in eradicating chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:- adequate organ function

* normal bone marrow cytogenetics Exclusion Criteria:- active CNS disease
* For autologous patients more than 30% bone marrow involvement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 1996-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Feasibility
Toxicity
olymerase Chain Reaction (PCR) for minimal residual disease

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Negrin, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States